CLINICAL TRIAL: NCT02257788
Title: PRO 140 2103: A Phase 2a, Randomized Study of PRO 140 by Subcutaneous Injection in Adult Subjects With Human Immunodeficiency Virus Type 1 Infection
Brief Title: PRO 140 for Human Immunodeficiency Virus Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unlikely to achieve targeted accrual
Sponsor: Drexel University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1210001606; 5U01AI095085-03 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Arm 1 (Active Comparator): PRO 140: one SC dose, 350 mg (day 1), followed by two single SC doses, 350 mg each (days 8 and 15) Intervention: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
  Interventions: Biological: PRO 140
- Treatment Arm 2 (Active Comparator): PRO 140: one SC loading dose, 700 mg (day 1), followed by two single SC doses, 350 mg each (days 8 and 15) Intervention: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
  Interventions: Biological: PRO 140
- Treatment Arm 3 (Active Comparator): PRO 140: one SC loading dose, 700 mg (day 1), followed by one single SC dose 350 mg (day 15) Intervention: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
  Interventions: Biological: PRO 140
- Treatment Arm 4 (Active Comparator): PRO 140: one SC dose, 700 mg (day 1) Intervention: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
  Interventions: Biological: PRO 140

INTERVENTIONS:
Biological: PRO 140 — Humanized monoclonal antibody to CCR5

SUMMARY:
PRO 140 2103 is a multicenter, randomized parallel group study, conducted in male and female adult subjects infected with CCR5-tropic HIV-1.

DETAILED DESCRIPTION:
Protocol PRO 140 2103 is a multicenter, randomized parallel group study, conducted in approximately 40 male and female adult subjects (n=10/treatment group) infected with CCR5-tropic HIV-1. Subjects will be randomized into one of four treatment groups. Blood samples for drug concentrations, PD variables, and efficacy variables will be obtained over a 59-day period following initiation of dosing. Safety will be monitored throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years
2. Has not taken any antiretroviral therapy (ART) within 12 weeks of the early screening visit
3. Screening plasma HIV-1 RNA ≥ 5,000 copies/mL
4. CD4+ lymphocyte cell count ≥500 cells/mm3 and no documented count less than or equal to 250 cells/mm3
5. Exclusive CCR5-tropic virus as determined by as determined by the Enhanced Sensitivity Trofile™ HIV Tropism Assay
6. Clinically normal resting 12-lead ECG at screening visit
7. Women of reproductive potential must have a negative serum pregnancy test at Late Screening Visit. Within hours prior to receiving the first dose of study drug, women of reproductive potential must have a negative urine pregnancy test. Male and female subjects must agree not to participate in a conception process and agree to use one barrier method of contraception plus one other highly reliable contraceptive method from the early screening visit through three weeks after the last administered subcutaneous dose of PRO 140.

Exclusion Criteria:

1. CXCR4-tropic virus, dual/mixed tropic (R5X4) virus as determined by the Enhanced Sensitivity Trofile™ HIV Tropism Assay
2. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
3. Diagnosis of acute viral hepatitis (defined as any active infection with hepatitis A or a new diagnosis of hepatitis B or C within 24 weeks of dosing)
4. Chronic hepatitis
5. Prior use of any entry, attachment, CCR5 coreceptor, or fusion inhibitor, including PRO 140, experimental or approved
6. Any immunization or vaccination (including influenza vaccine) within 30 days prior to administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum change in viral load following initiation of different dosing regimens of PRO140 | 59 days
  Viral Load is Defined as HIV-1 Copies/mL and Expressed as log10 Copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jacobson, MD, Study Chair — Drexel University
Locations (7):
- United States (7):
  - Stanford University (Stanford AIDS Clinical Trials Unit), Stanford, California
  - University of Colorado Denver (Colorado ACTU), Denver, Colorado
  - Washington University in St. Louis, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston (Houston AIDS Research team (HART), Houston, Texas